CLINICAL TRIAL: NCT07118878
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study to Assess Safety, Tolerability, and Pharmacokinetics of AGMB-129 in Healthy Participants
Brief Title: A Multiple Ascending Dose Study With AGMB-129 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agomab Spain S.L.U. (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: AGMB129-01-CL-109; 2025-521705-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-28; First posted 2025-08-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Fibrostenotic Crohn's Disease
Keywords: FSCD

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, double-blind, placebo-controlled, single-center study to evaluate the safety, tolerability, and PK of MADs of orally administered AGMB-129 compared with placebo in healthy participants.
  The study will evaluate up to 4 dose cohorts: 1 reference cohort with the reference dose of AGMB-129 BID and up to 3 MAD cohorts, including an optional cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, investigator(s), blinded monitors, and employees of the site involved in the management of the study will be blinded to intervention, unless in case of emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGMB-129 (Experimental): participants will receive a single dose of AGMB-129 (reference cohort) for 7 consecutive days or multiple doses of AGMB-129 (cohort 1, 2, 3) for 7 consecutive days
  Interventions: Drug: AGMB-129
- Placebo (Placebo Comparator): participants will receive a single dose of placebo (reference cohort) for 7 consecutive days or multiple doses of placebo (cohort 1, 2, 3) for 7 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AGMB-129 — AGMB-129
  Arms: AGMB-129
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In patients with Crohn's disease (CD), fibrosis of the gastrointestinal (GI) tract can result in stricture (stenosis) formation and obstruction of the GI tract, causing obstructive symptoms and often requiring surgical intervention. There are currently no approved therapies for treating fibrostenotic Crohn's disease (FSCD) and therefore, there is an urgent need for safe and effective antifibrotic therapies.

AGMB-129 has shown to be safe in healthy participants with single doses up to 1200 mg and multiple doses up to 200 mg twice daily (BID) for 10 days, and in FSCD patients with multiple doses up to 200 mg BID for 12 weeks.

This Phase 1 study will explore the safety, tolerability, and pharmacokinetics (PK) of other daily doses of AGMB-129 in healthy participants to inform on dose selection (nominal dose and dosing frequency) for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 55 years of age (extremes included), at the time of signing the informed consent.
2. Body weight of at least 50.0 kg for men and 45.0 kg for women, and a BMI between 19.0 and 30.0 kg/m2 (extremes included) at screening.
3. Male or female

Exclusion Criteria:

1. Known hypersensitivity to AGMB-129 ingredients or history of a significant allergic reaction to AGMB-129 ingredients as determined by the investigator.
2. Positive serology for HBsAg or anti-HCV antibodies at screening, or history of hepatitis from any cause except for hepatitis A that was resolved at least 3 months prior to the first administration of study treatment.
3. History of or a current immunosuppressive condition, including a positive test for HIV-1 or HIV-2 antibodies at screening.
4. Presence or sequelae of gastrointestinal, liver, kidney (eGFR ≤80 mL/min/1.73 m² using the CKD-EPI formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs at screening. Note: Participants who have an eGFR of up to 10% below 80 mL/min/1.73 m2 may be enrolled in the study at the discretion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Number of participant with Adverse Events | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of adverse events (AE) at every visit
Number of participant with abnormal Physical examination | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of physical examination at every visit
Number of participant with abnormal Vital signs | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of vital signs
Number of participant with abnormal electrocardiograms (ECGs) parameters | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal electrocardiograms (ECGs) at every visit
Number of participant with abnormal 2-dimensional (2-D) echocardiography | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal 2-dimensional (2-D) echocardiography at every visit
Number of participant with abnormal clinical laboratory tests | From enrollment to the end of treatment at 42 days
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal clinical laboratory parameters at every visit

SECONDARY OUTCOMES:
Plasma levels of AGMB-129 | From enrollment to the end of treatment at 42 days
  To characterize the pharmacokinetics (PK) of AGMB-129 by measuring the amount in plasma
Plasma levels of metabolite MET-158 | From enrollment to the end of treatment at 42 days
  To characterize the pharmacokinetics (PK) of metabolite MET-158 by measuring the amount in plasma
Plasma levels of metabolite MET-154 | From enrollment to the end of treatment at 42 days
  To characterize the pharmacokinetics (PK) of metabolite MET-158 by measuring the amount in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Fleurinck, MD, Study Director — Agomab Spain SL
Locations (1):
- SGS Belgium, Edegem, Belgium